CLINICAL TRIAL: NCT03057080
Title: Peripheral Angioplasty as the First Choice Revascularization Procedure to Promote Ischemic Leg Ulcer Healing
Brief Title: The Role of Percutaneous Angioplasty in Ischemic Leg Ulcer Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, MD, PhD, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTA1A
Record Dates: First submitted 2017-02-12; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Foot Ulcers
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTA procedure (Other): Percutaneous transluminal angioplasty (PTA) in patients with ischemic leg ulcer
  Interventions: Procedure: Percutaneous transluminal angioplasty (PTA)

INTERVENTIONS:
Procedure: Percutaneous transluminal angioplasty (PTA) — The main goal of the angioplasty (which was also the definition of technical success) was to achieve straight-line flow (SLF) from the aorta down to either a patent dorsalis pedis or plantar arch.

SUMMARY:
The aim of our study was to evaluate the technical and clinical effectiveness of PTA in the management of ischemic foot ulcers. All consecutive patients presenting with a foot ulcer at the outpatient Vascular surgery clinic of our hospital were evaluated. If non-invasive parameters suggested peripheral arterial disease (PAD) anatomic imaging (CTA and/or DSA) was performed and a PTA was carried out when feasible during the same session. All patients were followed until healing, amputation, death, or for at least two years. Short-term and long-term clinical success of PTA was evaluated based on ulcer size and appearance. Patients with worsening ulcers after PTA underwent bypass grafting or amputation.

DETAILED DESCRIPTION:
The aim of our study was to evaluate the technical and clinical effectiveness of PTA in the management of ischemic foot ulcers.

Methods: All consecutive patients presenting with a foot ulcer at the outpatient Vascular surgery clinic of our hospital were evaluated. Preoperative evaluation included foot pulse assessment, ankle-brachial-index (ABI) and duplex scanning. If non-invasive parameters suggested peripheral arterial disease (PAD) anatomic imaging (CTA and/or DSA) was performed and a PTA was carried out when feasible during the same session. All patients were followed until healing, amputation, death, or for at least two years. Short-term and long-term clinical success of PTA was evaluated based on ulcer size and appearance. Patients with worsening ulcers after PTA underwent bypass grafting or amputation.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed patients with ischemic foot ulcer and
* patients aged 18 years or older.

Exclusion Criteria:

* refusal to participate
* refusal of PTA therapy
* lesions not amenable to endovascular revascularization by vascular team's consensus based on preinterventional imaging
* absolute contraindication to contrast media injection, as determined by the investigator
* uncontrollable coagulopathy
* unwilling or unable to provide informed consent or return for required follow-up evaluations and
* previous or concurrent participation in another clinical research study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with ulcer healing | 2 years
  Number of patients with complete Ischemic leg ulcer healing defined as the complete epithelization of the lesion

SECONDARY OUTCOMES:
Amputation free survival | 2 years
  Number of months without amputation
Number of patients with all-cause mortality | 2 years
  Number of patients with all-cause mortality after PTA
Number of participants with Major adverse events | 2 years
  Number of participants with Major adverse events from PTA
Number of patients with 30-day morbidity and mortality | 30 days
  30-day morbidity and mortality from PTA
Number of patients requiring re-intervention | 2 years
  umber of patients requiring PTA re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tsetis, MD, PhD, Study Chair — University of Crete

IPD SHARING:
Plan to Share IPD: No